CLINICAL TRIAL: NCT07182162
Title: Development and Assessment of the Point-of-Care Ultrasound (PoCUS) Teleeducation Curriculum for Hospital-at-home Care: Using Near-Peer Training, Remote Supervision, and High-Fidelity Simulation
Brief Title: Point-of-Care Ultrasound (PoCUS) Teleeducation Curriculum for Hospital-at-home Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Attending physician, National Taiwan University Hospital, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 202501195RINB
Record Dates: First submitted 2025-09-11; First posted 2025-09-19 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-09

CONDITIONS: Educational Problems
Keywords: ultrasound; peer teaching; remote supervision; simulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote supervision + Simulation (Experimental): This group will experience didactics plus near-peer hands-on with remote supervision and scenario simulation (lecture + on-site near-peer instructor hands-on + simulation). The PoCUS teacher will not be physically present but will supervise remotely via video conferencing to monitor and communicate in real-time.
  Interventions: Other: Remote supervision + simulation
- Control (No Intervention): This group will follow the conventional teaching model, didactics plus on-site faculty-supervised hands-on (lecture + on-site teacher supervised hands-on).

INTERVENTIONS:
Other: Remote supervision + simulation — teacher use remote supervision to assist peer training Hospital-at-Home scenario simulation
  Arms: Remote supervision + Simulation

SUMMARY:
Since July 2024, the National Health Insurance Administration (NHIA) has been implementing a pilot Hospital-at-Home (HAH) Acute Care Program to curb hospital admissions. Point-of-Care Ultrasound (PoCUS) is considered the most promising imaging tool for this model. Replicating the hospital's familiar environment-its staffing patterns, diagnostic workflows, and medication protocols-in a patient's home or nursing facility is almost impossible, posing a major challenge to care teams. Medical-simulation training offers a solution, yet current PoCUS courses remain organ-based and lack scenario-based simulations that prepare physicians for HAH practice.

This two-year study will create a PoCUS curriculum and outcome-assessment tools tailored to HAH, adapting previously validated Entrustable Professional Activities (EPA) instruments to three HAH scenarios: pneumonia, urinary tract infection, and soft-tissue infection. Year 1 will develop scenario-based simulation courses and matching EPA tools, and train peer instructors who receive full PoCUS instruction for the three scenarios. Year 2 will randomly assign learners to compare two teaching models-peer training with remote supervision and scenario simulation versus traditional PoCUS training-evaluated with an Objective Structured Clinical Examination (OSCE) scored by EPA forms across multiple domains.

The project aims to establish normative standards for PoCUS training and assessment in HAH, confirm the feasibility of peer training with remote supervision, and provide a platform to train HAH medical teams nationwide, including those in rural areas.

DETAILED DESCRIPTION:
Background

PoCUS has evolved from hospital-based imaging to bedside diagnostic support, enabling rapid, problem-oriented assessments across trauma, shock, dyspnea, and resuscitation scenarios as portable devices matured in image quality and accessibility.

Recent medical education trends emphasize competency-based medical education (CBME), milestones, and EPAs, requiring structured assessment of indications, image acquisition, interpretation, and integration into management for skill-intensive technologies such as ultrasound.

Near-peer training can scale instruction without loss of effectiveness compared with faculty-led teaching, while remote supervision and simulation address logistical limits. However, online environments can attenuate nonverbal cues, underscoring the need for purposeful instructional design and validated evaluation tools.

Taiwan's National Health Insurance (NHI) launched a HAH pilot program in July 2024 focusing on acute infections-pneumonia, urinary tract infection (UTI), and soft tissue infection-where portable diagnostics and PoCUS can substitute or complement in-hospital imaging for timely home-based decisions.

Clinicians transitioning from hospital workflows to patients' homes and care facilities face new operational constraints, motivating scenario-based, high-fidelity simulation to rehearse dynamic conditions and multi-skill tasks that mirror real HAH care.

Objectives

The study aims to compare the effectiveness of a PoCUS curriculum using near-peer training with remote supervision and high-fidelity scenario simulation versus traditional on-site, in-person PoCUS teaching in the HAH context.

The study also aims to determine whether remote OSCE combined with EPA assessments are consistent with in-person evaluations and feasible for high-stakes skill appraisal. EPA-based assessment levels across four domains-Indication, Acquisition, Interpretation, and Integration-are anchored to OSCE cases aligned with HAH pneumonia, urinary tract infection, and soft tissue infection scenarios.

Methods

This is a two-year, prospective, randomized educational intervention study.

* Year 1: Development of HAH-focused scenario-based curricula; design of OSCE and EPA tools through expert consensus; and training of near-peer instructors who undergo rehearsal teaching with faculty observation and immediate feedback to qualify for Year 2 delivery roles.
* Year 2: Randomization of Post-Graduate Year (PGY) residents to receive either traditional PoCUS instruction (didactics plus on-site faculty-supervised hands-on training) or the new model (didactics plus near-peer hands-on training with remote supervision and scenario simulation). Outcomes will be measured by OSCE performance scored using EPA instruments.

Participants

The target population comprises PGY residents, internal medicine residents, and family medicine residents at National Taiwan University Hospital who volunteer to enroll, with a planned Year 2 sample size of approximately 100 participants.

Inclusion criteria are the above-mentioned residency trainees aged 20 years or older. Exclusion criteria include unwillingness to participate.

Outcomes

* Primary outcomes: Learning outcomes between traditional and near-peer training with remote supervision and simulation. Learning outcomes include self-assessment questionnaires and EPA-based OSCE scores.
* Secondary outcomes:

  1. Technology Acceptance Model (TAM) survey: Learners' feedback on the new curriculum, collected after the PoCUS course and before OSCE testing.
  2. OSCE survey: A post-OSCE survey on learner feedback regarding the examination itself.
  3. Inter-rater variability: Agreement between remote and in-person EPA-based OSCE ratings to establish feasibility and equivalence of the remote assessment tool.

ELIGIBILITY:
Inclusion Criteria:

■ PGY, internal medicine, and family medicine residents at National Taiwan University Hospital.

Exclusion Criteria:

■Unwillingness to participate in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
OSCE total and subscale scores on EPA-based PoCUS | 1 month
  The effectiveness of the curriculum will be evaluated approximately one month after completing the PoCUS course for both the experimental and control groups, using OSCE assessments incorporating EPA constructs. The OSCE will be evaluated independently by two reviewers(on site and remote), with the final score calculated as the average of their individual assessments. Students' performance will be analyzed based on their total OSCE scores as well as their scores for each construct of the EPA.

SECONDARY OUTCOMES:
Technology Acceptance Model (TAM) questionnaire total and subscale scores | 1 month
  Learners' feedback on the new curriculum, using the Technology Acceptance Model (TAM) will be collected after the PoCUS course and before the OSCE testing.
Post-OSCE survey score | 1 month
  After the OSCE, a survey on the feedback on OSCE test will also be conducted.
Inter-rater reliability of EPA-based OSCE ratings | 1 month
  Agreement between remote and in-person EPA-based OSCE ratings to establish feasibility and equivalence of this remote tool

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) regarding the survey of TAM model and feedbak on OSCE test will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: After publication of the study
Access Criteria: Upon request to the principal investigator with relevant IRB consent